CLINICAL TRIAL: NCT01624363
Title: Prevalence of Pancreatic Cysts During Routine EUS
Brief Title: Prevalence of Pancreatic Cysts During Routine Endoscopic Ultra Sound
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John DeWitt, Director, Endoscopic Ultrasound, Indiana University
Other Study IDs: 0906-23
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2016-08

CONDITIONS: Pancreatic Cysts
Keywords: Pancreatic cysts incidentally found during EUS
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing EUS: Patients undergoing EUS for non-pancreatic treatment.

SUMMARY:
The investigators are interested in performing a detailed examination of the pancreas via EUS (Endoscopic Ultra Sound)for patients referred for a non-pancreatic condition. The hypothesis is to make a statistical determination of how many pancreatic cysts the investigators discover incidentally.

DETAILED DESCRIPTION:
The prevalence of incidental pancreatic cysts discovered during EUS. (see data tables)

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria included: patients >18 years old with decision making capacity referred for EUS for any other indication other than the evaluation of a known pancreatic cyst, solid mass, or suspected mass.

Exclusion Criteria:

* Any known history or evidence of the following from any previous imaging study: pancreatic cyst, solid mass, suspected pancreatic mass, dilated main pancreatic duct
* Previous surgical resection of any portion of the upper GI tract such as Billroth II that would not permit complete EUS exam of the pancreas
* Laboratory and/or clinical evidence of ongoing acute pancreatitis
* Previous pancreatic surgical resection
* Pregnancy
* Incarceration
* High risk for sedation
* Coagulopathy and/or thrombocytopenia
* The patients underwent a complete EUS examination of the pancreas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were identified on the day of scheduled endoscopy.
Sampling Method: Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2009-09; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M. DeWitt, M.D., Principal Investigator — Indiana University
Locations (1):
- University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Results publication

REFERENCES:
- [Background] Sey MS, Teagarden S, Settles D, McGreevy K, Cote GA, Sherman S, McHenry L, LeBlanc JK, Al-Haddad M, DeWitt JM. Prospective Cross-Sectional Study of the Prevalence of Incidental Pancreatic Cysts During Routine Outpatient Endoscopic Ultrasound. Pancreas. 2015 Oct;44(7):1130-3. doi: 10.1097/MPA.0000000000000408. PMID 26335009

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Undergoing EUS: Patients undergoing EUS for non-pancreatic treatment.
  Diagnosis of a previously undetected pancreatic cyst: patients identified to have a pancreatic cyst, will need to be followed via imaging studies.
Period: Overall Study
Arm/Group | Patients Undergoing EUS
Started | 341
Completed | 341
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Undergoing EUS
Number analyzed (Participants) | 341
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 228
  >=65 years | 113
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187
  Male | 154
Region of Enrollment [Number; unit: participants]
  United States | 341

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Pancreatic Cysts During Routine EUS
Description: The purpose of this study is to identify the prevalence of pancreatic cysts in patients undergoing EUS for non-pancreatic indications .
Time Frame: 48 months
Measure: Median (95% Confidence Interval); unit: participants found to have a cyst
Units Other Than Participants: pancreas'
Arm/Group | Patients Undergoing EUS
Number analyzed (Participants) | 341
Number analyzed (pancreas') | 341
participants found to have a cyst | 46 [2 to 80]

ADVERSE EVENTS:
Time Frame: 48 months
Arm/Group | Patients Undergoing EUS
Serious Adverse Events (participants affected / at risk) | 0/341
Other Adverse Events (participants affected / at risk) | 0/314

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes